CLINICAL TRIAL: NCT00928265
Title: Safety and Efficacy of Neuroform3TM for Intracranial Aneurysm Treatment
Acronym: SENAT
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: SENAT
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial; stenting; endovascular treatment; stent-assisted coiling; cerebrovascular disease
MeSH Terms: conditions — Intracranial Aneurysm; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endovascular treatment of intracranial aneurysm. — Neuroform stent is used in conjunction of occlusives devices such as coils. Neuroform Stent allows the treatment of wide neck aneurysm with embolic coils. Put in front of the wide neck, it keeps the coils into the aneurysm and avoids them to fall in the parent artery, preventing coil protrusion.
  Accomplishes this by providing coil support at the neck of the aneurysm
  Other Names: Neuroform3TM Microdelivery Stent System; M003E3250100,M003E3250150,M003E3250200,; M003E3300100,M003E3300150,M003E3300200,M003E3300300; M003E3350100,M003E3350150,M003E3350200,M003E3350300; M003E3400100,M003E3400150,M003E400200,M003E400300; M003E3450100,M003E3450150,M003E3450200,M003E3450300

SUMMARY:
This is a prospective observational multicenter registry to evaluate safety and efficacy data on Neuroform3TM stenting for treatment with endovascular coiling of wide neck aneurysms on an intent to treat basis.

The objectives of this study are:

1. Assessment of morbidity-mortality at 1 month and 12-18 months following the treatment of the intracranial aneurysm with Neuroform3TM stent and endovascular coiling using the modified Rankin scale (mRS).
2. to evaluate adverse events.
3. Angiographic assessment at 12-18 months compared to the initial post-treatment assessment via the modified Raymond scale and same/better/worse scale.

DETAILED DESCRIPTION:
There is an increasing perception in the Neurovascular community - supported by extensive peer-to-peer and congress communications - that "stent-assisted coiling" of intracranial wide neck aneurysms improves the long term angiographic outcome of treated patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 year's old patient or above.
* every patient suffering from an un-ruptured or ruptured aneurysm, for whom the endovascular treatment approach using the Neuroform3TM stent is considered by the therapeutic team in charge.
* patient who has given his consent to participate to the study and to get his anonymized data collected

Exclusion Criteria:

* patient with dissecting or fusiform aneurysm
* treatment of several aneurysms in the same procedure, except adjacent aneurysm treated by the same stent
* severe vasospasm
* aneurysm associated with an arterio-venous malformation
* use of another Neuroform3TM stent
* woman pregnant or nursing
* patients not likely to be followed upon (living abroad)
* people protected by justice (safeguard of law, supervision or trusteeship)
* patient unsuitable to the anti-thrombotic and/or to anticoagulants therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient coming to the hospital to get an endovascular treatment of the aneurysm
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and Mortality associated with stenting and coiling | 30 days and 12-18 months post procedure
  Assessment of morbidity and mortality at 30 days and 12-18 months post endovascular treatment of wide neck aneurysm with a Neurform 3 stent and coiling as assessed by the modified Rankin scale (mRS).

SECONDARY OUTCOMES:
Efficacy of the Neuroform stent for treatment of wide neck aneurysms | post procedure and at 12-18 months post procedure
  Assessment of the morphological results post endovascular coiling and stenting of wide neck aneurysms and assessment of anatomical stability of the treatment at 12-18 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Biondi, Principal Investigator; Alain Bonafé, Principal Investigator
Locations (12):
- France (12):
  - Centre Hospitalier pellegrin, Bordeaux
  - CHU Hôpital de la Côte de Nacre, Caen
  - CHRU Salengro, Lille
  - CHU Limoges, Limoges
  - Hôpital Neurologique, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Nancy, Nancy
  - CHU Hôpital Guillaume et René Laënnec, Nantes
  - Hôpital Saint-Roch, Nice
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Fondation Rotschild, Paris

REFERENCES:
- [Background] International subarachnoid aneurysms trials. lancet 2003 feb,1;361 (9355):430-1
- [Background] Akpek S, Arat A, Morsi H, Klucznick RP, Strother CM, Mawad ME. Self-expandable stent-assisted coiling of wide-necked intracranial aneurysms: a single-center experience. AJNR Am J Neuroradiol. 2005 May;26(5):1223-31. PMID 15891189
- [Background] Alfke K, Straube T, Dorner L, Mehdorn HM, Jansen O. Treatment of intracranial broad-neck aneurysms with a new self-expanding stent and coil embolization. AJNR Am J Neuroradiol. 2004 Apr;25(4):584-91. PMID 15090346
- [Background] Barath K, Cassot F, Rufenacht DA, Fasel JH. Anatomically shaped internal carotid artery aneurysm in vitro model for flow analysis to evaluate stent effect. AJNR Am J Neuroradiol. 2004 Nov-Dec;25(10):1750-9. PMID 15569741
- [Background] Benitez RP, Silva MT, Klem J, Veznedaroglu E, Rosenwasser RH. Endovascular occlusion of wide-necked aneurysms with a new intracranial microstent (Neuroform) and detachable coils. Neurosurgery. 2004 Jun;54(6):1359-67; discussion 1368. doi: 10.1227/01.neu.0000124484.87635.cd. PMID 15157292
- [Background] Byrne JV, Bashiri M, Pasco A, Morris JH. A novel flexible endovascular stent for use in small and tortuous vessels. Neuroradiology. 2000 Jan;42(1):56-61. doi: 10.1007/s002340050015. PMID 10663475
- [Background] Canton G, Levy DI, Lasheras JC, Nelson PK. Flow changes caused by the sequential placement of stents across the neck of sidewall cerebral aneurysms. J Neurosurg. 2005 Nov;103(5):891-902. doi: 10.3171/jns.2005.103.5.0891. PMID 16304994
- [Background] dos Santos Souza MP, Agid R, Willinsky RA, Cusimano M, Montanera W, Wallace MC, terBrugge KG, Marotta TR. Microstent-assisted coiling for wide-necked intracranial aneurysms. Can J Neurol Sci. 2005 Feb;32(1):71-81. doi: 10.1017/s0317167100016917. PMID 15825550
- [Background] Fiorella D, Albuquerque FC, Han P, McDougall CG. Preliminary experience using the Neuroform stent for the treatment of cerebral aneurysms. Neurosurgery. 2004 Jan;54(1):6-16; discussion 16-7. doi: 10.1227/01.neu.0000097194.35781.ea. PMID 14683536
- [Background] Howington JU, Hanel RA, Harrigan MR, Levy EI, Guterman LR, Hopkins LN. The Neuroform stent, the first microcatheter-delivered stent for use in the intracranial circulation. Neurosurgery. 2004 Jan;54(1):2-5. doi: 10.1227/01.neu.0000099370.05758.4d. No abstract available. PMID 14683535
- [Background] Lylyk P, Ferrario A, Pasbon B, Miranda C, Doroszuk G. Buenos Aires experience with the Neuroform self-expanding stent for the treatment of intracranial aneurysms. J Neurosurg. 2005 Feb;102(2):235-41. doi: 10.3171/jns.2005.102.2.0235. PMID 15739550
- [Background] Murayama Y, Nien YL, Duckwiler G, Gobin YP, Jahan R, Frazee J, Martin N, Vinuela F. Guglielmi detachable coil embolization of cerebral aneurysms: 11 years' experience. J Neurosurg. 2003 May;98(5):959-66. doi: 10.3171/jns.2003.98.5.0959. PMID 12744354
- [Background] Wakhloo AK, Lanzino G, Lieber BB, Hopkins LN. Stents for intracranial aneurysms: the beginning of a new endovascular era? Neurosurgery. 1998 Aug;43(2):377-9. doi: 10.1097/00006123-199808000-00126. No abstract available. PMID 9696095